CLINICAL TRIAL: NCT01591018
Title: Risk Reduction of Symptomatic and Silent Brain Infarctions During Cardiac Surgery Due to Ultrasound Activation of Endogenous Fibrinolytic System Using Transcranial Doppler Monitoring
Brief Title: SONOlysis in Risk REduction of Symptomatic and Silent Brain infarCtions dUring Cardiac surgEry
Acronym: SONORESCUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Palacky University (Other); Ministry of Health, Czech Republic (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NT13498-4/2012
Record Dates: First submitted 2012-04-23; First posted 2012-05-03 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Bypass Graft Redo; Heart Valve Diseases
Keywords: sonolysis, brain infarction, prevention, cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases; Brain Infarction | interventions — Cardiac Surgical Procedures; Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cardiac surgery with sonolysis (Experimental): cardiac surgery (CABG or heart valve surgery) with sonolysis (continual transcranial Doppler monitoring)
  Interventions: Procedure: sonolysis; Procedure: cardiac surgery
- cardiac surgery without sonolysis (Placebo Comparator): cardiac surgery (CABG or heart valve surgery) without sonolysis (continual transcranial Doppler monitoring)
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Procedure: sonolysis — continual transcranial Doppler monitoring with max. diagnostic intensity for min. 60 minutes
  Other Names: sonothrombolysis; sonothrombotripsy
  Arms: cardiac surgery with sonolysis
Procedure: cardiac surgery — coronary artery bypass graft (CABG) heart valve replacement
  Other Names: coronary artery bypass graft (CABG); heart valve replacement

SUMMARY:
The aim of the project is to demonstrate a fibrinolytic effect of sonothrombolysis (continual transcranial Doppler monitoring) using 2 MHz diagnostic probe on the reduction of risk of brain infarctions due to the activation of endogenous fibrinolytic system during cardiac surgery (CS). 120 patients indicated for CS (CABG or valve replacement) will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions detected using MRI examination 24 hours after CEA or CS in 5% level of significance. Patients will be randomized - subgroup 1 will undergo a 40-240minute non-diagnostic TCD monitoring during CS, subgroup 2 will undergo interventions without TCD monitoring.

The aim of the project is a concordance with the aim No 1 of the Resort Program of a Research and Development: "Improvement of quality of life of patients using the modern therapeutic methods but with relative small positive effect of quality of life". The aim of the project is in concordance with a priority of announced public grant competition: "Development of the new therapeutic methods of cardiovascular disorders, especially coronary heart disease and stroke". Confirmation of our hypothesis that sonothrombolysis is able to activate endogenous fibrinolytic system during CS with consecutive reduction of the number and volume of brain infarcts, can lead to the increase of the safety of CS in patients. We can presume that up to 50% of patients indicated for CS can be treated using these methods in the future.

DETAILED DESCRIPTION:
AIM OF THE PROJECT The aim of the project is to demonstrate an effect of continual TCD monitoring using 2 MHz diagnostic probe with maximal diagnostic energy on the reduction of risk of brain microinfarctions due to the activation of endogenous fibrinolytic system and mechanical effect on emboli during CS.

The aim of the project is a concordance with the aim No 1 of the Resort program of a research and development in the years 2010-2015: "Improvement of quality of life of patients using the modern therapeutic methods but with relative small positive effect of quality of life". The aim of the project is in concordance with a priority of announced public grant competition: "Development of the new therapeutic methods of cardiovascular disorders, especially coronary heart disease and stroke".

HYPOTHESIS Sonothrombolysis lead to activation of fibrinolytic system in both healthy volunteers and acute stroke patients. In acute stroke patients, mechanical effect of sonothrombolysis is the second effect leading to acceleration of occluded artery recanalization. We hypothesize that combination of mechanical effect and activation of fibrinolytic system durin sonothrombolysis (TCD monitoring) during CS will lead to recanalization of small arterial occlusions caused by microembolization during intervention. The result will be reduction of volume and the number of brain infarctions in the territory of the monitored MCA.

120 patients indicated for CS will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions in the territory of athe monitored MCA detected using MRI examination 24 hours after CS in 5% level of statistical significance. Patients will be randomized into 2 subgroups. Subgroup 1 will undergo non-diagnostic TCD monitoring during CS. Subgroup 2 will undergo CS without TCD monitoring.

PATIENTS AND METHODS Patients: 120 patients indicated for CS (isolated coronary artery bypass surgery or isolated heart valve surgery) will be enrolled into the study during a 3-year period. All 120 patients will be randomized for standard CS and TCD monitored CS.

Clinical examinations: Physical and neurological examinations including evaluating of neurological impairment of neurological deficit in NIHSS scale, modified Rankin scale and cognitive testing (Mini Mental State Examination, Clock drawing test) will be performed before and 24 - 72 hours after CS.

Randomization: Randomization using computer generated random allocation will be used, separately for coronary artery bypass surgery and valve surgery patients.

Sonothrombolysis: In patients randomized into sonothrombolysis subgroup, MCA segment in depth 55 mm will be monitored for 40 - 240 minutes using a diagnostic 2 MHz probe with maximal diagnostic energy. Non-diagnostic TCD monitoring will be performed without detection of microembolic signals or detection of changes in blood flow. The second (control) subgroup will undergo a standard CS without sonothrombolysis.

MRI protocol will consists of 4 sequences: 1. Localizer; 2. T2TSE; 3. FLAIR; 4. DWI. Sequences 1-3 will be applied in the same level, they will have the same slice thickness and the same cut number. The slice thickness comprises its own cut thickness (5 mm) + distant factor (30%). Standard number of slices is 19. Standard slice level is considered to be a modified level of skull base due to the minimalization of distant artifacts EPI sequence. T2TSE: TR=4000/TE=99/ETL=9, FOV 230, FOV ph. 75%, matrix 256x256. FLAIR: 8050/112/ETL=21/2 conc., FOV 230, FOV ph. 76,6%, matrix 256x151. EPI-DWI: 4200/139/EPI f.=96/6 av., FOV 230, FOV ph. 100%, phase enc. direction A-P, matrix 128x96 with interpolation, phase partial Fourier 6/8, Bw 1346 Hz/Px, echo spacing 0.83 ms, TA. Sequence called "trace" with three types of MR pictures in every slice: (a) T2*EPI b=0; (b) DWI b=500; (c) DWI b=1000. The fourth type of images automatically created an ADC map (in-line postprocessing). DWI show a middle (average) diffusivity of every point of examined brain tissue when b value is 500 and 1000. This sequence is applied in order to assess hemorrhage (T2*EPI) and monitor sites of reduced diffusion (DWI, b=500 and 1000). New infarctions will be evaluated only in the territory of treated ICA.

Adverse effects: All adverse effects during 1 month after UM will be registered, especially all causes for new admissions to the hospital, worsening of neurological symptoms (>4 points in NIH stroke scale), brain edema, symptomatic and asymptomatic intracranial bleeding detected in control brain MRI.

Study protocol has been approved by the Ethics Committees in accordance with the principles and guidelines of the Declaration of Helsinki, 1975.

ELIGIBILITY:
Inclusion Criteria:

* age 40-90 years,
* sufficient temporal bone window for TCD with detectable blood flow in MCA,
* independent patient (modified Rankin score 0-2),
* informed consent signed by the patient,
* CS will be performed as an elective surgery with an extracorporeal circulation

Exclusion Criteria:

* contra-indication for MRI examination (pace-maker, implanted metal material, claustrophobia),
* emergent surgery,
* acute myocardial infarction,
* combined cardiac surgery,
* combined cardiac and carotid surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skoloudik D, Hurtikova E, Brat R, Herzig R; SONORESCUE Trial Group. Sonolysis in Prevention of Brain Infarction During Cardiac Surgery (SONORESCUE): Randomized, Controlled Trial. Medicine (Baltimore). 2016 May;95(20):e3615. doi: 10.1097/MD.0000000000003615. PMID 27196464
- See also: University Hospital Ostrava — http://fno.cz
- See also: Ministry of Health of Czech Republic — http://mzcr.cz

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In total, 120 of 214 screened patients fulfilled the inclusion criteria. Subjects were allocated to the sonolysis or control group randomly and equally.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.5 [61 to 71] | 69.0 [64 to 73] | 68 [62 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 37 | 32 | 69
Arterial Hypertension [Number; unit: participants]
  Participants with Arterial Hypertension | 48 | 47 | 95
  Participants without Arterial Hypertension | 12 | 13 | 25
Diabetes Mellitus [Number; unit: participants]
  Participants with Arterial Hypertension | 23 | 19 | 42
  Participants without Arterial Hypertension | 37 | 41 | 78
Hyperlipidemia [Number; unit: participants]
  Participants with Hyperlipidemia | 33 | 38 | 71
  Participants without Hyperlipidemia | 27 | 22 | 49
Coronary Heart Disease [Number; unit: participants]
  Participants with Coronary Heart Disease | 42 | 40 | 82
  Participants without Coronary Heart Disease | 18 | 20 | 38
Myocardial Infarction in History [Number; unit: participants]
  Participants with Myocardial Infarction | 14 | 12 | 26
  Participants without Myocardial Inf.arction | 46 | 48 | 94
Atrial Fibrillation [Number; unit: participants]
  Participants with Atrial Fibrillation | 33 | 30 | 63
  Participants without Atrial Fibrillation | 27 | 30 | 57
Transient Ischemic Attack (TIA) or Stroke [Number; unit: participants]
  Participants with TIA or Stroke | 3 | 3 | 6
  Participants without TIA or Stroke | 57 | 57 | 114
Smoking [Number; unit: participants]
  Smokers | 6 | 6 | 12
  Non-smokers | 54 | 54 | 108
Alcohol abuse [Number; unit: participants]
  Alcohol Abuse Participants | 1 | 0 | 1
  Abstinent or Social Drinker Participants | 59 | 60 | 119
Internal carotid artery (ICA) stenosis ≥ 50% [Number; unit: participants]
  Participants with ICA Stenosis | 6 | 4 | 10
  Participants without ICA Stenosis | 54 | 56 | 110
Type of surgery [Number; unit: participants]
  Coronary Artery Bypass Graft | 31 | 29 | 60
  Valve Surgery | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number od Participants With New Brain Infarction in the Monitored MCA Territory Detected Using MRI
Description: to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions and brain infarctions > 0.5 cm3 in the monitored MCA territory in sonolysis group detected using MRI examination 24 hours after cardiac surgery in 5% level of statistical significance
Time Frame: 24 hours after intervention
Measure: Number; unit: participants
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis
Number analyzed (Participants) | 60 | 60
participants
  Participants with new infraction | 8 | 16
  Participants without new infraction | 52 | 44
Statistical Analysis 1: Comparison: Cardiac Surgery With Sonolysis vs Cardiac Surgery Without Sonolysis; Sample size was based on an expected 20% reduction of new ischemic lesions on DW-MRI in the sonolysis group (estimated prevalence, 10%) compared with the control group (estimated prevalence, 30%); Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected — Pre-study calculations using chi-square test with a continuity correction showed that ≥60 patients in each group were needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8

2. Secondary Outcome: Cognitive Decline
Description: To demonstrate an effect of sonolysis on the reduction of cognitive decline after cardiac surgery measured by Adenbook´s Cognitive Examination - revised (ACE-R)ACE-R. Adenbook´s Cognitive Examination - revised (ACE-R) can aquire value 0 to 100. Higher value represents better cognitive functions.
Time Frame: 30 days after intervention
Population: 50 out of 60 participants completed all cognitive tests in cardiac surgery with sonolysis group.
  50 out of 60 participants completed all cognitive tests in cardiac surgery without sonolysis group.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis
Number analyzed (Participants) | 50 | 50
units on a scale | 80 [74 to 85] | 82 [76 to 87]

3. Secondary Outcome: Number of Participants With Clinical Manifested Brain Infarction
Description: to demonstrate an effect of sonolysis on the reduction of risk of clinically stroke due to the activation of endogenous fibrinolytic system during cardiac surgery
Time Frame: 30 days after intervention
Population: All enrolled participants were analyzed
Measure: Number; unit: participants
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis
Number analyzed (Participants) | 60 | 60
participants
  Participants with clinical manifested infarction | 0 | 2
  Participants without clinical manifest. infarction | 60 | 58

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Serious adverse events.
Arm/Group | Cardiac Surgery With Sonolysis | Cardiac Surgery Without Sonolysis
Serious Adverse Events (participants affected / at risk) | 42/60 | 44/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac Surgery With Sonolysis (N=60) | Cardiac Surgery Without Sonolysis (N=60)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Infection of respiratory system (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 24 (24)
Other infections (Infections and infestations) | 10 (12) | 11 (14)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Gastrointestinal disease (Gastrointestinal disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes